CLINICAL TRIAL: NCT02755298
Title: Chronic Clinical Effect of Acetazolamide in Pulmonary Hypertension
Brief Title: Chronic Clinical Effect of Acetazolamide
Acronym: ChronicAZA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KEK-ZH-2016-00089-2
Record Dates: First submitted 2016-03-24; First posted 2016-04-28 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Hypertension, Pulmonary
Keywords: Treatment Outcome; Acetazolamide
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetazolamide (Experimental): Twice a day 250 mg acetazolamide for 5 weeks
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo capsule 250 mg (Mannitol) twice a day 5 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide
  Arms: Acetazolamide
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study seeks primarily to determine the chronic clinical effect of AZA on exercise capacity (6MWD) compared to placebo.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) of various etiologies causes dyspnea, impairs exercise performance and is associated with reduced quality of life (QoL) and survival. Treatment options include therapy for any underlying causes, pulmonary vasodilator drugs, oxygen and, in selected cases, pulmonary endarterectomy or lung transplantation. Unfortunately, PH specific drugs are expensive, associated with side effects and even combined pharmacological treatment is often not sufficient to achieve clinical benefits. Therefore, novel therapeutic drugs are needed. We have recently demonstrated that sleep related breathing disorders, which are common in PH patients, can be improved by both nocturnal oxygen therapy and acetazolamide (AZA). AZA is a carbonic anhydrase (CA) inhibitor that acts as a respiratory stimulant thereby improving oxygenation and possibly PH. There are even data suggesting that CA-inhibitors have a direct pulmonary vasodilator effect. However, the potential role of AZA in the treatment of PH has not been conclusively studied. Therefore, the purpose of the current project is to investigate, the chronic clinical effects of AZA in PH patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing right heart catheterisation (RHC) for a clinical indication and who are diagnosed with precapillary PH (mean pulmonary arterial pressure (mPAP) ≥25 mmHg, pulmonary wedge pressure (PAWP) ≤15mmHg)
* Patients have to be in a stable condition, on the same medication for >4 weeks

Exclusion Criteria:

* Patients in whom a RHC is clinically not indicated
* pregnant women
* PH in left heart disease or with more than mild chronic obstructive pulmonary disease or restrictive lung disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Difference in 6 min walk distance | 5 weeks
  At the end of both periods (AZA and Placebo)

SECONDARY OUTCOMES:
Difference of Quality of Life (QoL) assessed by the physical subscale of the living with pulmonary hypertension questionnaire (MLHF) | 5 weeks
  At the end of both periods (AZA and Placebo)
Progressive maximal ramp cardiopulmonary exercise testing | 5 weeks
  At the end of both periods (AZA and Placebo)
cerebral and muscle tissue oxygenation | 5 weeks
  At the end of both periods (AZA and Placebo) at rest and exercise
daily activity | 5 weeks
  actigraphy
morphological and functional parameters of the heart | 5 weeks
  measured by echocardiography
New York Heart Association functional class | 5 weeks
  At the end of both periods (AZA and Placebo)
Short-form medical outcome questionnaire (SF-36) | 5 weeks
  At the end of both periods (AZA and Placebo)
Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) | 5 weeks
  At the end of both periods (AZA and Placebo)
N-terminal pro-brain natriuretic Peptide (NT-proBNP) | 5 weeks
  At the end of both periods (AZA and Placebo)
mean nocturnal oxygen Saturation during ambulatory sleep studies | 5 weeks
  At the end of both periods (AZA and Placebo)
apnea/hypopnea index during ambulatory sleep studies | 5 weeks
  At the end of both periods (AZA and Placebo)
Stroop test of cognitive performance | 5 weeks
  At the end of both periods (AZA and Placebo)
Trail making test (test of cognitive Performance) | 5 weeks
  At the end of both periods (AZA and Placebo)
5 point test (test of cognitive Performance) | 5 weeks
  At the end of both periods (AZA and Placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, MD, Principal Investigator — UniversityHospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lichtblau M, Saxer S, Muller J, Appenzeller P, Berlier C, Schneider SR, Mayer L, Furian M, Schwarz EI, Swenson ER, Bloch KE, Ulrich S. Effect of 5 weeks of oral acetazolamide on patients with pulmonary vascular disease: A randomized, double-blind, cross-over trial. Pulmonology. 2024 Jul-Aug;30(4):362-369. doi: 10.1016/j.pulmoe.2022.11.004. Epub 2023 Jan 11. PMID 36639329